CLINICAL TRIAL: NCT04610086
Title: Shared Decision Making and Satisfaction With the Diagnostic-therapeutic Process in the Context of the Colorectal Cancer Screening Program. The CyDESA Study.
Brief Title: Shared Decision Making and Satisfaction With the Diagnostic-therapeutic Process in the Shared Decision Making and Satisfaction With Colorectal Cancer Screening. The CyDESA Study
Acronym: CyDESA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Anna Selva, Medical Doctor, Corporacion Parc Tauli
Other Study IDs: PI18/00460
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer; Satisfaction, Patient
MeSH Terms: conditions — Colorectal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- False positive FIT: Participants in the colorectal cancer screening program, with a positive FIT and with a normal colonoscopy
- Polyps: Participants in the colorectal cancer screening program, with a positive FIT and diagnosed of colorectal polyps in the colonoscopy
- Colorectal cancer: Participants in the colorectal cancer screening program, with a positive FIT diagnosed by colorectal cancer

SUMMARY:
A cross sectional multicenter study (3 centers) to know the participation in decision making and the experience and satisfaction of participants with a positive immunological fecal test (FIT) result in relation to the screening process and the diagnostic-therapeutic process of cancer.

We will include 850 participants with a positive FIT result and will classify them by their final diagnosis (false positives of FIT; polyps; colo-rectal cancer).

Outcomes of interest will be measured by auto administered questionnaires:

collaboRATE, SDM-Q-9, OUT-PATSAT35 and a satisfaction questionnaire developed in a previous study.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the colorectal cancer screening program, with a positive result in the FIT AND in whom the perform of a colonoscopy is indicated AND agree to be included

Exclusion Criteria:

* People for whom the performance of a colonoscopy is not indicated by medical reasons
* People who refuse to perform a colonoscopy
* People who do not understand Spanish or Catalan, with deterioration of the cognitive state that do not allow them to understand or answer the questionnaires on their own or with the help of a caregiver;
* People in which the process is not carried out completely in the study centers (eg. performance of the colonoscopy in a private center).

Ages: 49 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participans in the colorectal cancer screening program with a positive results in the immunological fecal test.
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-02-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Satisfaction | Once the screening process is finished
  Satisfaction with the colorectal cancer screening programm

SECONDARY OUTCOMES:
Participation in decision making | Once the screening process is finished
  Patient perception of participation in decision making during the screening process
Satisfaction with diagnosis and treatment of cancer | at 6 months
  Satisfaction with the diagnostic and treatment processess of cancer
Participation in cancer decision making | at 6 months
  Patient perception about participation in decision making during the diagnostic and treatment processess of cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selva A, Lopez P, Puig T, Macia F, Selva C, Alvarez-Perez Y, Terraza R, Buron A, Machlab ST, Pericay C, Sola I, Tora N, Rodriguez V, Barrufet C, Aymar A, Bare M. Patient experience, satisfaction and shared decision-making in colorectal cancer screening: protocol of the mixed-methods study CyDESA. BMJ Open. 2022 May 30;12(5):e057687. doi: 10.1136/bmjopen-2021-057687. PMID 35636783